CLINICAL TRIAL: NCT04311788
Title: Preemer Trial - Prophylactic Mesh Versus no Mesh in the Midline Emergency Laparotomy Closure for Prevention of Incisional Hernia: a Multi Center, Double-blind, Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Elisa Mäkäräinen, Principal Investigator, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3/2020
Record Dates: First submitted 2020-03-07; First posted 2020-03-17 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Incisional Hernia; Emergency Laparotomy; Midline Laparotomy; Hernia Prevention
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Prophylactic self gripping mesh (Program, Medtronic) will be placed in rectorectus space to prevent incisional hernia.
  Interventions: Device: Prophylactic self gripping mesh
- Control group (Active Comparator): Abdomen of the patients in the control group will be closed by using small stitch closure with suture to wound length of 4:1 and slowly absorbable monofilament suture.
  Interventions: Device: Slowly absorbable continuous monofilament suture

INTERVENTIONS:
Device: Prophylactic self gripping mesh — Prophylactic self gripping mesh, Propgrip by Medtronic.
  Arms: Intervention group
Device: Slowly absorbable continuous monofilament suture — Fascial closure by continuous slowly absorbable 4:1 suture
  Arms: Control group

SUMMARY:
244 patients, who have an emergency midline laparotomy for any gastrointestinal reason, will be randomized in a 1:1 ratio either to mesh group with a retrorectus prophylactic self-gripping mesh or to control group with 4:1 small stitch closure by continuous monofilament suture. They will be followed up at 30 days, 2 and 5 years to detect the incidence of incisional hernia.

DETAILED DESCRIPTION:
Incisional hernia (IH) is a common complication of abdominal wall surgery. Its' incidence varies greatly (2-30 %) among studies. The incisional hernia incidence is influenced by several factors, such as closing technique, follow-up time and the modality of radiological investigations, patient characteristics and co-morbidities as well as indication and type for surgery.

European Hernia Society (EHS) guideline strongly recommends to utilise a non-midline approach to a laparotomy whenever possible to decrease the incidence of incisional hernia. However, this is clearly not an option in an emergency laparotomy, as midline incision is the fastest and the best visualizing opening to explore the whole abdominal cavity in an emergency setting.

For elective midline incisions, evidence-based recommendation is to perform a continuous suturing technique with slowly absorbable monofilament suture when closing the incision. Suturation should be done performing a single layer aponeurotic closure technique without separate closure of the peritoneum. A small bites technique with a suture to wound length (SL/WL) ratio at least 4:1 is the current recommended method of fascial closure.

Prophylactic mesh augmentation in a non-emergency setting appears effective and safe and can be suggested for high-risk patients. However, no recommendations can be given on the optimal technique to close emergency laparotomy incisions because of lack of evidence. This problem should be emphasized on due to high rates of IH after emergency laparotomy. All this makes the use of prophylactic mesh in the emergency setting an interesting proposition, as it may decrease the rate of IHs. However, there are concerns over potential mesh related complications including infection, chronic pain, seromas and bowel fistulas especially in emergency situations like peritonitis and intestinal obstruction. There is preliminary evidence published about the safety and efficiency of the prevention of IHs using meshes in the emergency laparotomy closure even in contaminated conditions.

In the resent systematic review and meta-analysis, only results of 2 studies and altogether 299 patients were eligible for the analysis. Swiss case-control study reported an IH rate of 3,2% (2/63) in the mesh group and 28,6% (20/70) in the control group. Spanish study group had the same kind of results in their retrospective cohort; IH rate of 5,9% (3/50) in the mesh group and 33,3% (33/100) in the control group. There was no statistically significant difference in the incidence of surgical site infection or other complications when prophylactic mesh group was compared to standard closure group. SSI rate in Swiss study was 60% and respectively only 17% in the Spanish study. This may reflect differences in the patient selection, therefore the safety profile of the prophylactic mesh in the emergency setting has not been adequately described. Neither of the studies included in meta-analysis were not randomized controlled trials. There were also many methodological differences including patient selection, used mesh, and mesh placement. Thus, the conclusion of the systematic review paper was that there are limited data to assess the effect or safety of the use of prophylactic mesh in the emergency laparotomy setting. Randomized control trials are required to address this important clinical question. EHS guideline group resulted the same conclusion in their recommendation report.

There are about 1650 patients are operated in Finland because of IH every year. According to the European study, the estimated cost for IH surgery is 6450 euros. The corresponding costs in Sweden were even higher reaching 9060 euros per treatment. Extrapolated to Finland, this means that operative treatment of IHs cause more than 10 million expenses to the Finnish health care sector in a year. Some of these costs may be avoidable by using the prophylactic mesh during the closure of midline emergency laparotomies in the patients with IH risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Midline emergency laparotomy for any gastrointestinal indication

Exclusion Criteria:

* • Previous ventral hernia repair with mesh in the midline

  * Previous inguinal or femoral hernia repair by any technique with mesh is accepted

    * Previous WHO class of physical activity 3-4 (WHO 3 more than 50% of time at rest, WHO 4 stays at rest most of the time)
    * Relaparotomy
    * Indication for laparotomy is incarcerated hernia
    * Pregnant or suspected pregnancy
    * <18 years
    * Metastastic malignancy of any origin
    * Planned osteomyelitis
    * Patients living geographically distant and/or unwilling to return for follow-ups
    * No informed consent
    * Subject participates in another RCT Intra-operative exclusion criteria applicable for both randomization groups
    * Abdomen is left open
    * Second look laparotomy planned
    * Ostomy created at the operation
    * Inability to keep the mesh securely out of the peritoneal cavity or close the anterior fascia
    * Intra-abdominal malignancy diagnosed at the operation
    * >2 cm hernia in midline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2025-02-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of incisional hernia | 2 years
  Incidence of incisional hernia, either symptomatic or asymptomatic detected clinically and/or radiologically

SECONDARY OUTCOMES:
Comprehensive Complication Index | 30 days
  Comprehensive Complication Index
Surgical site infection (SSI) rate | 30 days
  Surgical site infection (SSI) rate defined by CDC classification of surgical site infection
Fascial rupture | 30 days
  Incidence of fascial rupture
Incisional hernia | 5 years
  Incisional hernia incidence during long-term follow-up
Incisional hernia repair rate | 5 years
  Incisional hernia repair rate during follow-up
Re-operations | 5 years
  Re-operations due to mesh- or hernia related indications
Quality of life by RAND-36 | 5 years
  Quality of life defined by RAND-36
Quality of life by Promis | 5 years
  Quality of life defined by Promis questionnaire
Quality of life by AAS | 5 years
  Quality of life defined by AAS questionnaire
Cost analysis | 5 years
  All differences in costs between the groups will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Mäkäräinen-Uhlbäck, M.D., Principal Investigator — Oulu University Hospital
Locations (7):
- Finland (7):
  - Jorvi Hospital, Espoo
  - Helsinki University Hospital, Helsinki
  - Lahti Central Hospital, Lahti
  - Oulu University Hospital, Oulu
  - Seinäjoki Central Hospital, Seinäjoki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Makarainen E, Tolonen M, Sallinen V, Mentula P, Leppaniemi A, Ahonen M, Saarnio J, Pinta T, Lampela H, Malmi H, Lietzen E, Nikki M, Ohtonen P, Muysoms F, Rautio T. Prophylactic Retrorectus Mesh Versus Small-Stitch Closure After Emergency Midline Laparotomy: 2-Year Results of a Randomized Controlled Trial. J Abdom Wall Surg. 2025 Nov 27;4:15500. doi: 10.3389/jaws.2025.15500. eCollection 2025. PMID 41394095
- [Derived] Makarainen E, Tolonen M, Sallinen V, Mentula P, Leppaniemi A, Ahonen-Siirtola M, Saarnio J, Ohtonen P, Muysoms F, Rautio T. Prophylactic retrorectus mesh versus no mesh in midline emergency laparotomy closure for prevention of incisional hernia (PREEMER): study protocol for a multicentre, double-blinded, randomized controlled trial. BJS Open. 2022 Jan 6;6(1):zrab142. doi: 10.1093/bjsopen/zrab142. PMID 35143628

DOCUMENTS (1):
  • Study Protocol (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT04311788/Prot_000.pdf